CLINICAL TRIAL: NCT05482932
Title: The Numbers Tell the Tale: the Validation of an Assessment Battery for Health-related Physical Fitness in Patients with Inflammatory Bowel Disease
Brief Title: Health-related Physical Fitness in Patients with Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Gastroenterology & Hepatology Foundation (Maag Lever Darm Stichting) (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL79305.068.22; ZP 21-13 (Other Grant/Funding Number: Dutch Gastroenterology & Hepatology Foundation)
Record Dates: First submitted 2022-07-19; First posted 2022-08-01 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: Inflammatory bowel disease; Ulcerative Colitis; Crohn Disease; Health-related physical fitness
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with IBD: 100 patients with IBD; either Ulcerative Colitis (N=50) or Crohns disease (N=50)
  Interventions: Diagnostic Test: Health-related physical fitness assessment
- Healthy volunteers without IBD: 100 healthy volunteers (without IBD)
  Interventions: Diagnostic Test: Health-related physical fitness assessment

INTERVENTIONS:
Diagnostic Test: Health-related physical fitness assessment — Participants will complete several questionnaires and perform multiple health-related physical fitness tests

SUMMARY:
Rationale: Existing literature suggests an impaired health-related physical fitness (HRPF) (i.e., body composition, aerobic capacity, muscular strength, muscular endurance, and flexibility) in patients with inflammatory bowel disease (IBD). However, previous studies did not assess HRPF with the 5- component multidimensional concept. HRPF is not routinely screened for and measured within the IBD population in clinical practice. The lack of a simple screening tool and assessment method for HRPF validated for the IBD population hinders the ability to distinguish patients with IBD with adequate physical fitness from those who might benefit from physical exercise interventions targeting specific components. Gold standard measures are too expensive and too complex to implement in daily practice and therefore a screening tool and a simpler assessment battery for HRPF validated in patients with IBD are needed. It is necessary to obtain more objective insights into the specific components of HRPF affected in patients with IBD, and its association with patient-, disease-, and treatment-related factors in order to implement systematic screening in routine care and subsequently offer tailored physical exercise interventions.

Objective: The main objective of this study is to validate a simple screening tool and a best-practice assessment battery for the different components of HRPF against gold standard measures. Secondary objectives are to objectively assess the incidence of specific components affected in patients with IBD compared to healthy control subjects and to explore the association between these components of HRPF affected and patient-, disease-, and treatment-related factors.

DETAILED DESCRIPTION:
The study involves one or two study visits for patients with IBD and only one study visit for healthy volunteers. During the first study visit, all participants (n=200) will perform the tests of the assessment battery for HRPF and complete several questionnaires. A representative subgroup of patients with IBD will undergo the gold standard measurements for HRPF during a second study visit. Furthermore, total physical activity measured by accelerometry will be measured in this subgroup of patients.

ELIGIBILITY:
Inclusion criteria for all participants:

* Any gender aged 18 years or older;
* American Society of Anesthesiologists (ASA) Physical Status I or II (i.e., normal healthy patient or a patient with mild systemic disease)
* No contraindications for exercise testing based on the PAR-Q
* Being able to provide written informed consent;
* Willing and able to complete questionnaires and perform performance tests;
* Being able to understand written Dutch and speak the Dutch language.

Inclusion criteria specific for patients with IBD:

* Certified diagnosis of IBD (UC or CD) based on the combination of endoscopic, radiological, and/or histological findings;
* No active disease or experiencing mild to moderate disease activity.
* Included in eHealth clinical care-pathway using myIBDcoach.

Inclusion criteria specific for healthy volunteers:

• No certified diagnosis of IBD (CD, UC, IBD-Unclassified);

Exclusion criteria for all participants:

* ASA Physical Status > II (i.e., patient with severe systemic disease);
* Contraindications for exercise testing based on PAR-Q
* Other (temporary) injuries or severe (neuro)muscular, rheumatic, or orthopedic conditions that may interfere with study evaluations;
* Current malignancy (except for local cutaneous skin cancer) or successfully treated for a malignancy in the past 6 months;
* Pregnant or lactating women;
* Competitive and elite athletes (i.e., ≥6 hours/week of moderate to vigorous exercise)
* Not being able to understand or speak the Dutch language;
* Not being able to cooperate with test procedures or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with IBD will be recruited at the gastroenterology outpatient clinic of the Maastricht UMC+. Healthy volunteers will be recruited by means of advertisements in publicly accessible sites such as the hospital, university, and social media, as well as via advertisements as posters in the hospital and university.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-09-27 (Actual)

PRIMARY OUTCOMES:
Duke Activity Status Index | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: estimated VO2peak
Veterans-Specific Activity Questionnaire | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: estimated METs
Sum of 4 skinfold thicknessess | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: % body fat, fat mass, fat free mass
Bioelectrical impedance analysis | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: % body fat, fat mass, fat free mass
Mid upper arm circumference | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: cm
Waist circumference | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: cm
Steep ramp test (peak work rate) | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: peak work rate
Handgrip strength | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: kg
Handgrip endurance | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: seconds to task failure (sec)
Handheld dynamometry | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: peak torque
1 minute sit-to-stand test | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: repetitions
sit-and-reach test | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: cm
Deuterium oxide dilution (Only applicable for first 50 included patients with IBD) | Study visit 2, 7 to 14 days after inclusion (cross sectional study design)
  Outcome: % body fat, fat mass, fat free mass).
Cardiopulmonary exercise test (Only applicable for first 50 included patients with IBD) | Study visit 2, 7 to 14 days after inclusion (cross sectional study design)
  Outcome: VO2max/VO2peak)
Biodex 4 Pro dynamometry (Only applicable for first 50 included patients with IBD) | Study visit 2, 7 to 14 days after inclusion (cross sectional study design)
  Outcome: peak torque

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: MET min/week
Total physical activity measured with accelerometer (Only applicable for first 50 included patients with IBD) | 7 days (between 1st and 2nd study visit)
  Outcome: total physical activity, number of steps and intensity, time spent in posture and intensity
Checklist Individual Strength | Study visit 1, at time of inclusion (cross sectional study design)
  Outcome: fatigue

OTHER OUTCOMES:
Patient characteristics | At time of inclusion (cross sectional study design)
  e.g., age, gender, medical history, comorbidities, IBD phenotype, disease duration, extra-intestinal manifestation, medication use, tobacco use

CONTACTS AND LOCATIONS:
Overall Officials: M.J. Pierik, Prof., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center +, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided